CLINICAL TRIAL: NCT00002362
Title: A Randomized, Open-Label Superiority Trial Comparing Emtricitabine to Abacavir Within a Triple Drug Combination in Antiretroviral-Drug Naive HIV-1 Infected Patients
Brief Title: A Comparison of Emtricitabine and Abacavir Used in a Three-Drug Combination in HIV-Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: Triangle Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 298B; FTC-301
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-03

CONDITIONS: HIV Infections
Keywords: Dideoxynucleosides; Drug Therapy, Combination; Stavudine; Reverse Transcriptase Inhibitors; abacavir; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — abacavir; efavirenz; Emtricitabine; Stavudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Efavirenz
Drug: Emtricitabine
Drug: Stavudine

SUMMARY:
This study will look at whether emtricitabine is as safe and effective as abacavir (ABC) when taken with stavudine (d4T) and efavirenz (EFV) in patients who have never taken anti-HIV drugs.

DETAILED DESCRIPTION:
Patients are randomized to receive open-label emtricitabine or ABC in combination with stavudine and efavirenz. Viral load and CD4+ cell counts are compared at Weeks 24 and 48. Patients are followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

You may be eligible if you:

* Are HIV-positive and generally healthy.
* Have a viral load of 5,000 copies/ml or more.
* Have CD4 cell counts of 200 cells/mm3 or more.
* Are age 18 or older.
* Agree to practice sexual abstinence or use effective barrier methods of birth control (such as condoms).

Exclusion Criteria

You will not be eligible if you:

* Have ever taken anti-HIV drugs for 3 days or more.
* Have had certain AIDS-related infections.
* Have had severe diarrhea within the past 30 days.
* Are unable to eat at least 1 meal a day due to nausea, vomiting, or stomach pain.
* Are being treated for active tuberculosis (TB).
* Are pregnant or breast-feeding.
* Use illegal drugs or alcohol that make it difficult for you to take study drugs or keep clinic appointments.
* Are taking certain medications, or have certain other conditions or diseases (see the technical summary for more detail).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Ctr for AIDS Research / Education and Service (CARES), Sacramento, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Gary Richmond MD, Fort Lauderdale, Florida
  - Northstar Med Clinic, Chicago, Illinois
  - South Jersey Infectious Diseases Inc, Somers Point, New Jersey
  - North Shore Univ Hosp / Div of Infectious Diseases, Manhasset, New York
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Univ of Texas / Med School at Houston, Houston, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas